CLINICAL TRIAL: NCT06433973
Title: Comparative Evaluation of Root Coverage Outcome by Using CM With Photobiostimulation ,CM & SCTG in Treating Isolated RT 2 Recession Defects Utilizing Minimally Invasive Technique: A RCT
Brief Title: Chorion Membrane With Photobiostimulation ,Chorion Membrane & SCTG in Treating Isolated RT 2 Recession Defects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anisha Kumari Perio 24/36
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1 - CM+LLLT+VISTA (Experimental): After obtaining adequate LA exposed root surfaces of treated teeth are to be scaled with curettes to reduce root convexity and undercuts.CM will be placed on the recession defect using minimally invasive technique. Photobiostimulation will be done using of diode laser.
  Interventions: Procedure: Test group 1 - CM+LLLT+VISTA
- Test group 2 - CM+VISTA (Experimental): After obtaining adequate LA exposed root surfaces of treated teeth are to be scaled with curettes to reduce root convexity and undercuts.CM will be placed on the recession defect using minimally invasive technique.
  Interventions: Procedure: Test group 2 - CM+VISTA
- Control group - SCTG+VISTA (Other): Scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage procedure will be done with CTG using minimally invasive access technique.
  Interventions: Procedure: Control group - SCTG+VISTA

INTERVENTIONS:
Procedure: Test group 1 - CM+LLLT+VISTA — After obtaining adequate LA exposed root surfaces of treated teeth are to be scaled with curettes to reduce root convexity and undercuts.CM will be placed on the recession defect using minimally invasive technique. LLLT will be applied on the site for 10 sec.
  Arms: Test group 1 - CM+LLLT+VISTA
Procedure: Test group 2 - CM+VISTA — After obtaining adequate LA exposed root surfaces of treated teeth are to be scaled with curettes to reduce root convexity and undercuts. Adequate size of CM will be trimmed and applied over the recession defect using minimally invasive technique and secured with sutures.
  Arms: Test group 2 - CM+VISTA
Procedure: Control group - SCTG+VISTA — Scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage procedure will be done with CTG using minimally invasive access technique.
  Arms: Control group - SCTG+VISTA

SUMMARY:
Gingival recession (GR) is defined as apical displacement of the gingival margin relative to the cemento-enamel junction, with resultant oral exposure of the root.

Most of the recessions in periodontal patients involve the destruction of interproximal periodontal tissues, and these were classifed as Miller class III and IV or Cairo RT2 andRT3 gingival recessions (GRs).

Taking all this into account, numerous techniques have been attempted to achieve root coverage of single-rooted tooth, Connective tissue graft presently stands as the benchmark in periodontal plastic surgery, offering excellent predictability and enhanced long-term root coverage. However, its availability is limited and its use often leads to increased patient morbidity.Thus making placental allografts in dentistry a topic of growing interest and recent advancement.

It may be hypothesized that CM + LLLT or CM may be used an alternative to SCTG in minimally invasive technique in recession coverage. Hence, this study evaluates root coverage percentages in RT2 gingival defects using a CM with and without photobiostimulation, comparing them to each other and to SCTG- the gold standard control group.

DETAILED DESCRIPTION:
Most of the recessions in periodontal patients involve the destruction of interproximal periodontal tissues, therefore, these were classified as Miller class III and IV or Cairo RT2 and RT3 gingival recessions (GRs). The growing emphasis on aesthetics and the desire to minimize patient discomfort have led to the advancement of various mucogingival techniques aimed at covering exposed roots. numerous techniques have been attempted to achieve root coverage of single-rooted tooth. Connective tissue graft presently stands as the benchmark in periodontal plastic surgery, offering excellent predictability and enhanced long-term root coverage. However, its availability is limited and its use often leads to increased patient morbidity. Thus making placental allografts in dentistry a topic of growing interest and recent advancement. Other advantages like their capacity to self hydrate with blood. While these techniques have proven effective, the integration of devices capable of accelerating wound healing could enhance the outcomes of the latest graft techniques for root coverage, facilitating more predictable results.

Progress in low-level laser therapy (LLLT) within Periodontics has empowered periodontists to attain enhanced clinical outcomes. LLLT accelerates wound healing by enhancing the motility of human keratinocytes, stimulating early epithelialization, increasing fibroblast proliferation and matrix synthesis, and promoting neo vascularization.

.LLLT induces tissue surface sterilization, there by reducing the risk of bacteremia, and diminishing edema, swelling, and scarring .Additionally, it may provide greater tensile strength and stability to gingival margins, potentially preventing wound failure and reducing clinical recession. Besides all the advantages of LLLT and chorion membrane, there are very few studies which are published using theses two techniques in the recession defects. No prior research has examined the comparative efficacy of SCTG, CM + LLLT and CM for Miller's class III/RT2 recession defects. It may be hypothesized that CM + LLLT or CM may be used an alternative to SCTG in minimally invasive technique in recession coverage. Hence, this study evaluates root coverage percentages in RT2 gingival defects using a CM with and without photobiostimulation, comparing them to each other and to SCTG- the gold standard control group

ELIGIBILITY:
Inclusion Criteria:

* Patients with Millers class3or RT2 isolated recession defects in labial mandibular anterior teeth region.
* Systemically healthy individuals.
* Absence of clinical tooth mobility.
* Age >18 years old.
* A full mouth plaque index < 20%
* Patient showing adequate compliance and willing to participate in the study.

Exclusion Criteria:

* Patients having systemic disease such as hypertension, diabetes, hyperthyroidism or on medication that influence the outcome of periodontal therapy.
* patient with active periodontal disease
* smokers and tobacco users
* mal-alingned lower anteriors.
* patients who had already undergone root coverage procedure on the selected site.
* pregnant and lactating females
* Involved tooth with trauma from occlusion.
* Involved tooth with prosthesis.
* Endodontically involved/ RCT treated tooth
* Tooth with cervical abrasion / undetectable CEJ/ carious.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage root coverage | 6 months
  ( Preoperative recession depth) - (Postoperative recession depth) × 100
  Preoperative recession depth
Keratinised tissue width | 6 months
  recorded in mm with a periodontal probe, from the crest of gingival margin to the mucogingival junction.
interproximal Clinical attachment level (iCAL) | 6 months
  recorded in mm with a periodontal probe from the cemento enamel junction to the base of the pocket by inserting the periodontal probe at the interproximal region

SECONDARY OUTCOMES:
Bleeding on probing (BOP) | 6 months
  will be recorded as 1(present) if bleeding occurs within 15 seconds of probing and 0(absent) if no bleeding occurs. It will be calculated in percentage %. After adding all the scores, total score will be divided by the total number of surfaces accessed and multiplied by hundred. It will be designed as percentage sites with bleeding on probing
Buccal Clinical attachment level | 6 months
  recorded in mm with a periodontal probe from the cemento enamel junction to the base of the pocket by inserting the periodontal probe at the mid-buccal region
change in Gingival thickness | 6 months
  The GT will be assessed by probe transparency (TRAN) method
  . Gingival thickness will be measured from the keratinized mucosa to the periosteum with a finger spreader and a silicon slider and digital calliper at a point lying in the centre of a line drawn from the gingival margin to mucogingival junction
Recession depth | 6 months
  recorded in mm with a periodontal probe from the cementoenamel junction to the crest of the gingival margin at the mid-labial region.
Recession width | 6 months
  recorded in mm with a periodontal probe from the mesial to distal gingival margin at the level of cementoenamel junction
Pocket probing depth | 6 months
  Measured in mm from the crest of the gingival margin to the base of the pocket at the mid-labial region
Patient based evaluation of pain and hypersensitivity by visual analogue scale for pain(VAS) | 6 months
  The visual analogue scale (VAS) is considered to be one of the best methods available for the estimation of the intensity of pain. Postoperative pain using visual analog scale at treated site (VAS: a scale from 0-10 ; 0 means no pain/discomfort, 10 means maximum pain /discomfort )

CONTACTS AND LOCATIONS:
Overall Officials: Anisha Kumari, BDS, Principal Investigator — PGIDS, Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No